CLINICAL TRIAL: NCT02753621
Title: Parkinsonics: A Controlled Study of Group Singing for Quality of Life and Voice Outcomes in Parkinson Disease
Brief Title: Parkinsonics: A Controlled Study of Group Singing in Parkinson Disease
Acronym: Parkinsonics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Alex Pantelyat, Assistant Professor of Neurology, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00065196
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Singing Intervention (Experimental): Twelve weekly group singing classes lasting 60-90 minutes under the direction of a professional choir director and a social worker with a music background.
  Interventions: Behavioral: Group singing
- Discussion/Support Group Intervention (Active Comparator): Twelve weekly 60-90 minute discussion groups led by a facilitator trained in discussion group facilitation; occurring at the same time and in the same location (next door) as experimental intervention (group singing).
  Interventions: Behavioral: Facilitated Discussion Group

INTERVENTIONS:
Behavioral: Group singing — Weekly group singing classes led by professional choir instructor, lasting 90 minutes. 12 classes over 12 consecutive weeks.
  Arms: Singing Intervention
Behavioral: Facilitated Discussion Group — Weekly facilitated discussion group led by Parkinson Disease educator, lasting 90 minutes. 12 sessions over 12 consecutive weeks.
  Arms: Discussion/Support Group Intervention

SUMMARY:
The overall objective of this study is to observe the effect of group Vocal performance training and performance experience on patients' reported symptoms and quality of life. The effectiveness of PD medications varies significantly in different patients depending on their symptoms. By using music-based interventions to improve symptoms that may be inadequately treated by medications, the investigators hope to improve quality of life in PD patients. "Parkinsonics: A controlled study of group singing for quality of life and voice outcomes in Parkinson disease" (PD) is a controlled crossover behavioral intervention study of once weekly choral classes for patients with idiopathic PD (progressing toward a group performance) and once weekly discussion/support group meetings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD based on UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria for PD (Hughes et al. 1992).

Exclusion Criteria:

* Patients unable to consent to the study.
* Patients unable or unwilling to participate in weekly singing classes for 12 weeks, or unwilling to perform in a concert setting.
* Patients with active psychiatric disturbances (agitation, active hallucinations).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Parkinson Disease Quality of Life Questionnaire (PDQ)-39 scores | Change from baseline scores at 30 weeks
  Validated 39-item questionnaire

SECONDARY OUTCOMES:
Voice-Related Quality of Life | Change from baseline scores at 30 weeks
  Validated 10-item questionnaire
Movement Disorder Society-Unified Parkinson Disease Rating Scale Motor scores | Change from baseline scores at 30 weeks
  Validated Parkinson disease motor assessment scale
Montreal Cognitive Assessment | Change from baseline scores at 30 weeks
  Validated cognitive assessment
Geriatric Depression Scale-15 | Change from baseline scores at 30 weeks
  Validated depression self-rating
Lorig Self-efficacy scale | Change from baseline scores at 30 weeks
  5-item self-reported questionnaire
Short Form-36 | Change from baseline scores at 30 weeks
  Self-reported questionnaire assessing patients' health based on their physical and mental well-being
Sound pressure level (decibels) | Change from baseline levels at 30 weeks
  Assessed while reading the standardized "Rainbow" passage and describing the cookie theft picture at a 50cm distance from the microphone (using a portable professional decibel meter).
Voice jitter | Change from baseline values at 30 weeks
  Analysis will be performed using Praat software (Boersma and Weenink, version 5.4.01, http://www.fon.hum.uva.nl/praat/). There will be 3 trials per subject holding sounds A and E for as long as possible on one breath. Sound recordings are made for each trial.
Voice shimmer | Change from baseline values at 30 weeks
  Analysis will be performed using Praat software (Boersma and Weenink, version 5.4.01, http://www.fon.hum.uva.nl/praat/). There will be 3 trials per subject holding sounds A and E for as long as possible on one breath. Sound recordings are made for each trial.
Harmonic to noise ratio | Change from baseline values at 30 weeks
  Analysis will be performed using Praat software (Boersma and Weenink, version 5.4.01, http://www.fon.hum.uva.nl/praat/). There will be 3 trials per subject holding sounds A and E for as long as possible on one breath. Sound recordings are made for each trial.

OTHER OUTCOMES:
Feasibility | 12 weeks
  At least 80% of participants attending at least 9 of 12 singing classes and the final performance

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Pantelyat, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No